CLINICAL TRIAL: NCT06682741
Title: Comparison of the Effects of Different Training Programs on the Levels of Cognitive Function
Brief Title: Comparison of Different Training Programs on Cognitive Function
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 433/24
Record Dates: First submitted 2024-09-18; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: physical activity; neurotrophins; neuroprotection; cognitive function; MCI
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- excercise (Experimental): supervised exercise training; twice a week for 12 months
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — supervised exercise training; twice a week for 12 months

SUMMARY:
The goal of the project is to identify the most effective exercise modalities in terms of neuroprotective effects and FP improvement.

Hypothesis: Dancing will increase BDNF, GDNF and CLU levels to a greater extent than traditional forms of AF, resulting in significantly greater improvements in FP in subjects aged ≥ 60 years. The study will involve 60 women aged ≥ 60 years, randomly and equitably assigned to training groups (i.e., resistance training using body weight, dance) and a control group (i.e., a group of physically inactive women).

Methodology:

Participants: 60 women aged ≥ 60 randomly and equally assigned to training groups (Dance and Resistance training) and a control group (i.e., physically inactive women)

Scientists will compare the impact of different forms of physical activity on cognitive functions

DETAILED DESCRIPTION:
The training interventions will last 6 months. The intensity of physical activity will be determined as a percentage of maximum heart rate (HRmax), assessed based on a fitness test (Chester Step Test), using data from mobile devices monitoring physical activity. Cognitive function (CF) levels, and the concentrations of GDNF, BDNF, and CLU, as well as the Chester Step Test, will be evaluated twice: once at baseline and once after the training programs. Blood samples for measuring neurotrophin and CLU levels will be collected in the morning, after an overnight fast (approximately 12 hours since the last meal). The concentrations of neurotrophins and CLU will be measured using the ELISA method. CF will be assessed using standardized and validated neuropsychological tests.

Expected Outcomes: Greater improvement in CF in the dance group compared to the resistance training and control groups, with higher levels of BDNF, GDNF, and CLU in the dance group.

ELIGIBILITY:
Inclusion Criteria:

* women

Exclusion Criteria:

* previous diagnoses of cardiovascular diseases

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
tle level of cognitive functions | before and after 12 months of interventions
  Cognitive functioning is assessed using the standardized MoCA test, which has a maximum score of 30 points. A score of 26 or higher is considered normal

SECONDARY OUTCOMES:
blood markers | before and after 12 months of intervention
  Neurotrophins, such as BDNF (Brain-Derived Neurotrophic Factor) and GDNF (Glial-Derived Neurotrophic Factor), as well as clusterin are measured from blood using an ELISA test kit

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Ratajczak, PhD, Study Director — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Poland, Poland

IPD SHARING:
Plan to Share IPD: No